CLINICAL TRIAL: NCT06760858
Title: A Prospective Cohort Study on the Treatment of Locally Advanced Gastric Cancer with SOX Plus Tislelizumab Combined with HIPEC
Brief Title: A Prospective Cohort Study on the Treatment of Locally Advanced Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Yan Shi, Chief Physician, Southwest Hospital, China
Other Study IDs: SYIO-01
Record Dates: First submitted 2024-11-07; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer, Gastroesophageal Junction Cancer
Keywords: neoadjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab: 200mg IV, day 1, Q3W, for a total of 3 cycles.
Drug: SOX — SOX: S-1 dosage based on body surface area (BSA): <1.25m², 40 mg bid orally, 1.25-1.5m², 50 mg bid orally, ≥1.5m², 60mg bid orally, days 1-14; Q3W; Oxaliplatin 130mg/m² IV day 1, for a total of 3 cycles.
Device: HIPEC — HIPEC: Docetaxel: 120mg, day 1, day 3.

SUMMARY:
The clinical trial aims to assess the efficacy and safety of Tislelizumab combined with the SOX regimen and HIPEC in treating locally advanced gastric cancer. The primary and secondary objectives are as follows:

To evaluate the 3-year disease-free survival (DFS) in patients with locally advanced gastric cancer treated with systemic SOX chemotherapy plus Tislelizumab and HIPEC.

To assess the major pathological response (MPR) in these patients. Secondary objectives include safety, pathological complete response (pCR), progression-free survival (PFS), tumor regression grade (TRG), overall survival (OS), incidence of adverse reactions during treatment, postoperative adverse reactions, and treatment efficacy.

Participants will:

Be willing to receive SOX plus Tislelizumab combined with HIPEC treatment (exposure group), undergo HIPEC followed by SOX and Tislelizumab to achieve stable disease (SD), partial response (PR), or complete response (CR). Patients who can undergo surgery after the second exploration will receive surgery and HIPEC treatment. If surgery is not possible, a multidisciplinary team (MDT) discussion will follow to determine the next treatment plan. Patients with progressive disease (PD) will also have an MDT discussion to determine the subsequent treatment.

Be willing to receive SOX combined with HIPEC treatment (observation group), undergo HIPEC followed by SOX to achieve SD, PR, or CR. Patients who can undergo surgery after the second exploration will receive surgery and HIPEC treatment. If surgery is not possible, an MDT discussion will follow to determine the next treatment plan. Patients with PD will also have an MDT discussion to determine the subsequent treatment.

Treatment details:

SOX: S-1 dosage based on body surface area (BSA): <1.25m², 40 mg bid orally, 1.25-1.5m², 50 mg bid orally, ≥1.5m², 60mg bid orally, days 1-14; Q3W; Oxaliplatin 130mg/m² IV day 1, for a total of 3 cycles.

Tislelizumab: 200mg IV, day 1, Q3W, for a total of 3 cycles. HIPEC: Docetaxel: 120mg, day 1, day 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed Her-2 negative gastric adenocarcinoma, with no prior chemotherapy, radiotherapy, or other anti-cancer treatments before the start of the clinical trial.
* Age between 18 to 80 years old, Eastern Cooperative Oncology Group (ECOG) performance status: 0-1.
* Staging according to the American Joint Committee on Cancer (AJCC) 8th edition is T4aNxM0, without obstruction, perforation, or bleeding risk.
* Good bone marrow reserve function, with the following blood criteria: white blood cell count ≥3×10^9/L, neutrophils ≥1.5×10^9/L, platelet count ≥100×10^9/L, hemoglobin ≥90 g/L.
* Good organ function, with the following biochemical criteria: aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN), alanine aminotransferase (ALT) ≤2.5×ULN, serum total bilirubin ≤1.5×ULN, serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min.
* International normalized ratio (INR) ≤1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5 times ULN.
* Urine protein <2+, if urine protein ≥2+ then 24-hour urine protein quantification must be ≤1g.
* Consent to provide blood and tissue samples.
* Expected survival of more than 3 months.
* Female subjects agree to strict contraception; male subjects with partners of childbearing potential agree to use effective contraception during the study period.
* Voluntarily sign the informed consent form, willing and able to comply with planned visits, study treatments, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Participants who have been enrolled in any other drug clinical trial or have participated in any drug clinical trial within the last month.
* Any anti-cancer treatments (chemotherapy, radiotherapy, surgery, immunotherapy, biotherapy, chemoembolization) other than the study medication (palliative external beam radiation for non-target lesions is allowed).
* Prior use of similar chemotherapy drugs or immune checkpoint inhibitors.
* Presence of metastatic lesions in the liver, lungs, para-aortic lymph nodes, bones, brain, adrenal glands, or pelvic and abdominal cavity.
* Gastrointestinal perforation, obstruction, or uncontrollable diarrhea within 6 months prior to enrollment.
* Other untreated or concurrent tumors, except for cervical carcinoma in situ, treated basal cell carcinoma, or superficial bladder tumors. Patients with tumors that have been cured and have no evidence of disease for more than 5 years may be included. All other tumors must have been treated at least 5 years prior to enrollment.
* Symptomatic meningiomas：
* History of active autoimmune diseases or refractory autoimmune diseases.
* Received corticosteroids (>10mg/day prednisone or equivalent dose of steroids) or other systemic immunosuppressive therapy within 14 days prior to enrollment, excluding the following treatments: steroid hormone replacement therapy (≤10mg/day); local steroid therapy; and short-term prophylactic steroid therapy for allergies or nausea and vomiting.
* History of HIV infection or active hepatitis B/C virus infection.
* Persistent > Grade 2 bacterial, fungal, viral infections.
* Active or clinically significant cardiac disease:
* Congestive heart failure > New York Heart Association (NYHA) Class II;
* Active coronary artery disease;
* Arrhythmias requiring treatment other than beta-blockers or digoxin;
* Unstable angina (angina symptoms at rest), new-onset angina within 3 months prior to enrollment, or unhealed wounds, ulcers, or fractures due to myocardial infarction within 6 months prior to enrollment.
* Patients with renal failure requiring hemodialysis or peritoneal dialysis.
* Patients requiring medication for epilepsy.
* History of organ transplantation (including corneal transplants).
* Allergy to the study medication or similar drugs, or suspected allergies.
* Pregnant or breastfeeding women.
* Major surgery, open biopsy, or significant traumatic surgery within 4 weeks prior to recruitment.
* History of vaccination within 4 weeks prior to enrollment.
* Patients deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed Her-2 negative gastric adenocarcinoma，Staging according to the American Joint Committee on Cancer (AJCC) 8th edition is T4aNxM0, without obstruction, perforation, or bleeding risk
Sampling Method: Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years
  The 3-year disease-free survival (DFS) in patients with locally advanced gastric cancer treated with systemic SOX chemotherapy plus Tislelizumab combined with HIPEC

SECONDARY OUTCOMES:
MPR | 1 year
  Systemic SOX chemotherapy combined with Tislelizumab and HIPEC for locally advanced gastric cancer patients' major pathological response (MPR).

CONTACTS AND LOCATIONS:
Locations (1):
- The Southwest hospital of AMU, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No